CLINICAL TRIAL: NCT06899477
Title: Pre-Operative Treatment in REseCTable COlon CanceR (PROTECTOR/FIRE-10; AIO-KRK-0620; IAG-VO-0323) Prospective, Randomized, Open, Multicenter Phase III Trial to Investigate the Efficacy Preoperative Systemic Therapy in Advanced Colon Cancer
Brief Title: Pre-Operative Treatment in REseCTable COlon CanceR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dominik Paul Modest (Other)
Collaborators: Frankfurter Institut für Klinische Krebsforschung IKF GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Dominik Paul Modest, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROTECTOR/FIRE-10; 2023-508076-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Colo-rectal Cancer; Colon Cancer; Colon Carcinoma
Keywords: colo-rectal cancer; colon; neoadjuvant; upper rectum; pre-operative
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin; Oxaliplatin; Fluorouracil; Irinotecan

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open, multicenter Phase III trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Pre-operative treatment (Experimental): Arm A: choice of one of the offered pre-operative regimens:
  1. Up to 6 cycles, every 2 weeks, mFOLFOXIRI
  2. Up to 6 cycles, every 2 weeks, mFOLFOX-6
  3. Up to 4 cycles, every 3 weeks, CAPOX followed by structured Follow-up for up to 60months after randomization
  Interventions: Drug: mFOLFOXIRI; Drug: mFOLFOX-6; Drug: CAPOX
- Arm B: Control (No Intervention): Structured follow-up for at least 60 months after randomization

INTERVENTIONS:
Drug: mFOLFOXIRI — Up to 6 cycles, every 2 weeks, mFOLFOXIRI: Oxaliplatin 85 mg/m2 2 h day 1, Irinotecan 150 mg/m2 60-90 min day 1, Folinic acid 400 mg/m2 ~1 h day 1, followed by 5-FU 2400 mg/m2 46 h
  Other Names: Folinic acid, Oxaliplatin, 5-FU, Irinotecan
  Arms: Arm A: Pre-operative treatment
Drug: mFOLFOX-6 — Up to 6 cycles, every 2 weeks, mFOLFOX-6: Oxaliplatin 85 mg/m2 2 h day 1, Folinic acid 400 mg/m2 ~1 h day 1, (optional: 5-FU 400 mg/m2 bolus), followed by 5-FU 2400 mg/m2 46 h.
  Other Names: Folinic acid, Oxaliplatin, 5-fluorouracil (FU)
  Arms: Arm A: Pre-operative treatment
Drug: CAPOX — Up to 4 cycles, every 3 weeks, CAPOX: Oxaliplatin 130 mg/m2 3 h day 1, Capecitabine 1000 mg/m2 ORALLY taken twice daily d1-d14
  Other Names: Capecitaine, Oxaliplatin
  Arms: Arm A: Pre-operative treatment

SUMMARY:
This is an open-label, randomized, controlled, multicenter, phase III study with two parallel arms. Patients with advanced colon cancer, including the upper third of the rectum, clinically staged cT3-4 and or cN+ (defined as lymph nodes with short axis of at least 1cm) are randomized in a 2:1 fashion (favoring preoperative therapy= Arm A) to investigate the efficacy, patient reported quality of life and safety of preoperative mFOLFOXIRI or mFOLFOX-6 or CAPOX followed by surgery versus the standard of care algorithm (surgery followed by stage-guided adjuvant therapy as recommended by the local multidisciplinary tumor board (Arm B)).

DETAILED DESCRIPTION:
The trial will consist of a clinical and translational part. After completion of the treatment algorithm in both arms of the trial, follow-up as scheduled by current guidelines is recommended. Additionally, assessment of quality of life and blood sampling (tumor markers, circulating tumor DNA and potential innovative markers) will be performed for up to 5 years on a three-months basis. During the active part of the study, a radiologic re-assessment prior to surgery will be recommended for all trial subjects of arm A. Tumor biopsies and resected tumor specimens will be collected at screening (baseline sample) and in the course of treatment. Additionally, in case of disease relapse a tumor re-biopsy will be collected as far as considered feasible and safe for the patient by the investigator.

The objective of the re-assessments is detection of relapse either radiologically or within the translational material (blood samples with ctDNA dynamics and tumor - if available from relapses).

Patients in Arm A will receive a preoperative study drug intervention (mFOLFOXIRI or mFOLFOX-6 or CAPOX) for up to 3 months (6 cycles biweekly or 4 cycles triweekly) after randomization with clinical and safety assessments as specified in (Table 1).

Allocation to study treatment FOLFOX/FOLFOXIRI or CAPOX for patients in Arm A is stratified and done by investigator's choice. Beyond clinical or radiological factors, the decision may consider but is not limited to factors such as age, performance status, and patients' perspectives. Since obligatory criteria cannot be made, treatment allocation will not be regulated by the protocol, but stratification will avoid that treatment allocation promotes bias.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's signed informed consent.
2. Patient's age ≥18 years at the time of signing the informed consent.
3. Histologically confirmed adenocarcinoma of the colon or upper rectum.
4. Confirmed mismatch-repair proficient and/or microsatellite stable tumor. Both Immunohistochemistry and PCR can be used for diagnosis.
5. Intent for curative surgery
6. Predicted T3 or T4 stage and or nodal positivity (N+) in a computed tomography and/or magnetic resonance imaging scan of the abdomen/pelvis as assessed by the local study team.

   * T3-4 defined as invasion of surrounding tissue structures or organs
   * N+ defined as regional lymph node(s) without fat hilus and short axis diameter of ≥1 cm
7. Absence of clear distant metastases assessed by the investigator based on respective routine evaluations within 6 weeks prior to inclusion into the trial (preferred: computed tomography of thorax and abdomen. Alternatively magnetic resonance images, sonography and x-rays might be used for assessment).
8. Absence of significant active wound healing including severe chronic non-healing wounds, ulcerous lesions or untreated bone fracture
9. ECOG performance status 0-2.
10. Adequate bone marrow, hepatic and renal organ function, defined by the following laboratory test results:

    * Absolute neutrophil count ≥ 1.5 x 109/L (1,500/µL)
    * Hemoglobin ≥ 80 g/L (8 g/dL) with or without transfusion
    * Platelet count ≥ 100 x109/L (100,000/µL) without transfusion
    * Total serum bilirubin of ≤ 1.5 x upper limit of normal (ULN)
    * Aspartate aminotransferase (AST/GOT) ≤ 3.0 × ULN.
    * Calculated glomerular filtration rate (GFR) according to Cockcroft-Gault formula or according to MDRD ≥ 50 mL/min or serum creatinine ≤ 1.5 x ULN
11. Patients without anticoagulation need to present with an INR < 1.5 x ULN and PTT < 1.5 x ULN. Patient with prophylactic or therapeutic anticoagulation are allowed into the trial.
12. Proficient fluorouracil metabolism as defined:

    1. Prior treatment with 5-FU or capecitabine without unusal toxicity or
    2. If tested, normal DPD deficiency test according to the standard of the study site or
    3. If tested, in patients with DPD deficiency test with a CPIC activity score of 1.0-1.5 fluoropyrimidine dosage should be reduced by 50%
13. For women of childbearing potential (WOCBP): negative pregnancy test within 7 days before treatment initiation and agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study treatment.

A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male partner's sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

For men: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment. Men must refrain from donating sperm during this same period.

With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of study medication to avoid exposing the embryo.

Exclusion Criteria:

1. Ileus or directly imminent ileus as assessed by the local study team. Patients with treated and resolved ileus are allowed into the trial.
2. Previous chemotherapy for colorectal cancer of any stage
3. New York Heart Association Class III or greater heart failure by clinical judgement.
4. Myocardial infarction within 6 months prior to randomization; percutaneous transluminal coronary angioplasty (PTCA) with or without stenting within 6 months prior to randomization.
5. Unstable angina pectoris.
6. Unstable cardiac arrhythmia > grade 2 NCI CTCAE despite anti-arrhythmic therapy.
7. Ongoing toxicities > grade 2 NCI CTCAE, in particular peripheral neuropathy.
8. Active uncontrolled infection by investigator's perspective.
9. Known hypersensitivity to 5-FU, folinic acid, capecitabine, irinotecan or oxaliplatin or to any of the other excipients listed in section 6.1 of the corresponding SmPC.
10. Recent or concomitant treatment with brivudine.
11. Peripheral sensitive neuropathy with functional impairment (> grade 1 acc. to CTCAE version 5.0 (see appendix 2)).
12. Simultaneous application of St. John's Wort preparations.
13. Pernicious or other megaloblastic anemia caused by vitamin B12 deficiency.
14. Major surgical procedure, open biopsy, or significant traumatic injury within 21 days prior to randomization that may interfere with systemic therapy as judged by the investigator.
15. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications, including but not limited to:

    * Simultaneous application of live vaccines during treatment with irinotecan and for at least 6 months after the last dose.
    * 5-FU must not be given in combination with brivudin, sorivudin and analogues to patients homozygous for DPD and patients known with completely missing DPD activity.
    * Severe diarrhoea.
16. Medical history of malignant disease other than colorectal cancer with the following exceptions:

    * patients who have been disease-free for at least three years before randomization
    * patients with adequately treated and completely resected basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer, stage I uterine cancer
    * patients with any treated or untreated malignant disease that is associated with a 5-year survival prognosis of ≥ 90% and does not require active therapy
17. Known alcohol or drug abuse.
18. Pregnant or breastfeeding females.
19. Participation in a clinical trial or experimental drug treatment within 28 days prior to potential inclusion in the clinical trial or within a period of 5 half-lives of the substances administered in a clinical trial or during an experimental drug treatment prior to potential inclusion in the clinical trial, depending on which period is longest, or simultaneous participation in another clinical trial while taking part in this clinical trial.
20. Patients depended on Sponsor, investigator or study site.
21. Patient committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
22. Limited legal capacity

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2033-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | LPI + 36 months (96 months total)
  Disease-free survival (DFS) - defined as no surgery, no resection, incomplete resection, disease recurrence (new metastases or local relapse) and death from any cause from the time of randomization. In case of no surgery ,no resection, or incomplete resection (defined as R2 resection = macroscopic tumor rest), the timepoint of the respective event will be set to two weeks after randomization to avoid time-bias in favor of the experimental/neoadjuvant therapy arm.

SECONDARY OUTCOMES:
Overall survival (OS) | LPI + 60 months (120 months total)
  time from randomization to the date of death of any cause
Tumor regression grades (TRS) | LPI + 60 months (120 months total)
  according to Dworak's score
(Serious) Adverse Events | LPI + 60 months (120 months total)
  Type, incidence, severity, and causal relationship to active chemotherapy of non-serious adverse events and serious adverse events (severity evaluated according to CTCAE version 5.0), rate of surgery complication scores (Clavien Dindo)
Quality of life (QoL) | LPI + 60 months (120 months total)
  assessed with the QoL questionnaire EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Modest, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (28):
- Germany (28):
  - Charité Universitätsmedizin Berlin, Berlin
  - Ev. Waldkrankenhaus Spandau, Berlin-Spandau
  - Klinikum Chemnitz gGmbH, Chemnitz
  - St. Elisabeth Krankenhaus GmbH, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Gefos Dortmund mbH, Dortmund
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Hämatologisch Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - MediProject GbR, Hanover
  - St. Anna Hospital Herne, Herne
  - Sana Klinikum Hof, Hof
  - Alexianer Krefeld GmbH, Krefeld
  - ÜBAG MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - Gastroenterologie, Onkologie u. Diabetologie - Theresienkrankenhaus, Mannheim
  - GEHO, Münster
  - MVZ Media Vita, Münster
  - medius Klinik Ostfildern-Ruit, Ostfildern
  - Brüderkrankenhaus Sr. Josef, Paderborn
  - Kreiskliniken Reutlingen GmbH, Reutlingen
  - Mathias Spital - Klinikum Rheine, Rheine
  - RoMed Klinikum Rosenheim, Rosenheim
  - Leopoldina Krankenhaus, Schweinfurt
  - Marien Kliniken - St. Marienkrankenhaus Siegen, Siegen
  - MVZ Klinik Dr. Hancken GmbH, Stade
  - Lahn-Dill-Kliniken GmbH, Wetzlar
  - Remus-Murr-Kliniken gGmbH, Winnenden
  - Marien Hospital / MVZ, Witten

IPD SHARING:
Plan to Share IPD: No